CLINICAL TRIAL: NCT00095953
Title: A Phase II Study of SB-715992 (NSC 727990) in Previously Untreated Patients With Metastatic or Recurrent Malignant Melanoma
Brief Title: SB-715992 in Treating Patients With Metastatic or Recurrent Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I169; CAN-NCIC-IND169; CDR0000391842 (Other: PDQ)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2011-09

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — ispinesib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ispinesib — SB-715992 will be given as a 1 hour intravenous infusion in a dose of 18 mg/m2 once every 3 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as SB-715992, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well SB-715992 works in treating patients with metastatic or recurrent malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of SB-715992, in terms of response rate, in patients with previously untreated metastatic or recurrent malignant melanoma.
* Determine the toxic effects of this drug in these patients.
* Determine the early progression rate and response duration in patients treated with this drug.
* Determine the pharmacokinetics of this drug in these patients.
* Correlate pharmacokinetics with safety and efficacy endpoints of this drug in these patients.
* Correlate β-tubulin and kinesin spindle protein expression in tumor tissue with clinical outcomes in patients treated with this drug.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

All patients are followed at 4 weeks after completion of protocol therapy. Patients with ongoing complete response, partial response, or stable disease are followed every 3 months thereafter until relapse.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study within 12-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Previously untreated metastatic or recurrent disease
  * Considered incurable by standard therapies
* Measurable disease

  * At least one unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Bone metastases are not considered measurable disease
  * Outside any previously irradiated area

    * Patients whose sole site of measurable disease is in a previously irradiated area are ineligible unless there is evidence of progression or new lesions documented in the irradiated field
* No known CNS metastases

  * CT scans or MRI are not required to rule out CNS metastases unless patient exhibits neurological signs or symptoms
  * Patients with a prior solitary brain metastasis surgically resected with no evidence of residual disease are eligible provided CT scan or MRI confirms no evidence of disease within the past 28 days
* Archival paraffin tumor specimen available

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid tumors with no evidence of disease for ≥ 5 years
* No other uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to SB-715992

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior adjuvant immunotherapy
* No prior immunotherapy for metastatic or recurrent disease

Chemotherapy

* No prior chemotherapy, including regional therapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy except for low-dose, non-myelosuppressive radiotherapy

Surgery

* See Disease Characteristics
* At least 4 weeks since prior major surgery

Other

* More than 28 days since prior investigational agents
* More than 14 days since prior and no concurrent use of any of the following CYP3A4 inhibitors or inducers:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Itraconazole
  * Ketoconazole
  * Fluconazole (≤ 200 mg/day allowed)
  * Voriconazole
  * Nefazodone
  * Fluvoxamine
  * Verapamil
  * Diltiazem
  * Grapefruit juice
  * Bitter orange
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Oxcarbazepine
  * Rifampin
  * Rifabutin
  * Rifapentine
  * Hypericum perforatum (St. John's wort)
  * Modafinil
* At least 6 months since prior and no concurrent amiodarone
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer treatment
* No other concurrent investigational therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-11; Primary Completion 2006-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Response | 2 years

SECONDARY OUTCOMES:
Toxicity | 2 years
Pharmacokinetics at day 1 of course 1 (day 1 of course 2 if dose is changed) | 2 years
Molecular correlates on archival tissue, fresh tumor tissue, and peripheral blood mononuclear cells (PVMCs) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lee, MD, Study Chair — BCCA - Fraser Valley Cancer Centre
Locations (7):
- Canada (7):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - Nova Scotia Cancer Centre at Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Toronto Sunnybrook Regional Cancer Centre at Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

REFERENCES:
- [Result] Lee CW, Belanger K, Rao SC, Petrella TM, Tozer RG, Wood L, Savage KJ, Eisenhauer EA, Synold TW, Wainman N, Seymour L. A phase II study of ispinesib (SB-715992) in patients with metastatic or recurrent malignant melanoma: a National Cancer Institute of Canada Clinical Trials Group trial. Invest New Drugs. 2008 Jun;26(3):249-55. doi: 10.1007/s10637-007-9097-9. Epub 2007 Oct 26. PMID 17962907